CLINICAL TRIAL: NCT03225248
Title: Multi-center, Randomized, Active-Controlled, Double-Blind, Non-Inferiority, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of UI05MSP015CT in Functional Dyspepsia (MARS Study)
Brief Title: Efficacy and Safety of UI05MSP015CT in Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUP-MSP5-301
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UI05MSP015CT (Experimental): UI05MSP015CT and Placebo of Gasmotin
  Interventions: Drug: UI05MSP015CT
- Gasmotin (Active Comparator): Placebo of UI05MSP015CT and Gasmotin
  Interventions: Drug: Gasmotin

INTERVENTIONS:
Drug: UI05MSP015CT — UI05MSP015CT and Placebo of Gasmotin
  Arms: UI05MSP015CT
Drug: Gasmotin — Placebo of UI05MSP015CT and Gasmotin
  Arms: Gasmotin

SUMMARY:
This study is a multi-center, randomized, active-controlled, double-blind, non-inferiority, phase III clinical trial evaluating efficacy and safety of once-daily mosapride (UI05MSP015CT) in patients with functional dyspepsia.

DETAILED DESCRIPTION:
Patients with functional dyspepsia were randomly assigned (1:1) to receive either UI05MSP015CT (15 mg once daily before breakfast, study group) or mosapride (5 mg three times a day before each meal, control group) and corresponding placebo t.i.d. or q.d. for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age >19 years
2. Diagnosis of functional dyspepsia meeting Rome III criteria
3. At least three moderate or severe symptoms included in the Symptom Score
4. No structural lesions of upper gastrointestinal tract

Exclusion Criteria:

1. History of dyspepsia unrelated to functional dyspepsia or diseases
2. History of gastrointestinal surgery
3. History of malignancy in the previous 5 years
4. Psychiatric disorders including major depressive disorder and anxiety
5. Liver cirrhosis or abnormal liver laboratory findings
6. Advanced chronic kidney disease
7. Uncontrolled hypertension
8. Uncontrolled diabetes
9. Pregnancy and lactation
10. Recent history of taking medication affecting the gastrointestinal system

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2015-09-05 (Actual); Study Completion 2015-10-12 (Actual)

PRIMARY OUTCOMES:
Change of symptom score of functional dyspepsia | 4weeks
  Change of symptom score of functional dyspepsia was evaluated by symptom-specific questionnaire.

SECONDARY OUTCOMES:
Change of symptom score of functional dyspepsia | 2weeks
  Change of symptom score of functional dyspepsia was evaluated by symptom-specific questionnaire.
General symptom improvement | 2weeks, 4weeks
  Selecting: 'loss of symptom', 'apparent improvement', 'moderate improvement', 'no change', and 'deterioration'.
NDI-K questionnaire | 4weeks
  25 questions on five quality of life areas

IPD SHARING:
Plan to Share IPD: No